CLINICAL TRIAL: NCT07375836
Title: The Effect of Chocolate Consumption During Labor on Second Stage Duration
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0200-25-HYMC
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Labor; Second Stage of Labor; Pregnancy
Keywords: Second stage of labor; Oral carbohydrate intake; Non-pharmacologic intervention; Maternal exhaustion; Pregnancy; Labor; Randomized controlled trial

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel-group interventional study. Eligible participants will be randomized in a 1:1 ratio to receive either oral carbohydrate supplementation (chocolate) prior to second stage of labor, or standard intrapartum care. Outcomes will be compared between groups. The primary outcome is the duration of second stage of labor, with secondary maternal and neonatal outcomes assessed.
Masking Description: This is an open-label study. Masking is not feasible due to the nature of the intervention. However, the primary outcome is an objective measure, minimizing the risk of assessment bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 50 g of milk chocolate cocoa content 25-30% (Experimental): . Participants in the intervention group will receive one serving of 50 grams of milk chocolate (cocoa content 25-30%, without filling or additives) at a cervical dilation of 6 cm or more. The mother will be asked to consume the serving gradually over 30 minutes.
  Interventions: Other: 50 g of milk chocolate cocoa content 25-30%
- control group - no intervention (No Intervention): Participants in the control group will receive routine care as is customary in the delivery room, without any proactive nutritional supplementation.

INTERVENTIONS:
Other: 50 g of milk chocolate cocoa content 25-30% — Milk chocolate was chosen as it is better tolerated compared to dark chocolate, has a milder profile of active ingredients (which can increase nausea and heartburn) and provides a source of available carbohydrates.
  A dose of 50 grams was chosen that provides 25-30 grams of simple carbohydrates - sufficient for a significant increase in blood glucose but low enough to prevent a sudden sugar load or nausea.
  The intervention will be given at 6-9 cm dilation, towards the transition to the second phase - to allow the absorption of glucose and neurochemicals to be deafened at a time when the body needs increased energy and alertness. Giving it earlier may result in the effect of the chocolate wearing off before the second phase, and later - there will be no time for effective absorption.
  Arms: 50 g of milk chocolate cocoa content 25-30%

SUMMARY:
Childbirth is an energy-intensive physiological process, requiring sustained effort comparable in intensity to moderate physical activity. Studies suggest that providing an available energy source during labor, such as dextrose infusion or natural carbohydrate-rich foods such as dates, may shorten the duration of labor and improve cervical dilation without adversely affecting obstetric outcomes. The primary objective of the study is to examine whether giving chocolate during labor affects the duration of the second stage of labor, compared to a control group that will not receive a nutritional intervention. The study is a prospective, randomized, controlled trial that will be conducted in the delivery room of Hillel Yaffe Medical Center. Healthy pregnant women with a singleton pregnancy at ≥37 weeks gestational age, in spontaneous or induced labor, without diabetes (pre/gestational), will be recruited to participate. Participants in the intervention group will receive one serving of 50 grams of milk chocolate (cocoa content 25-30%, without filling or additives) at a cervical dilation of 6 cm or more (and not yet fully dilated). The mother will be asked to consume the serving gradually over 30 minutes. Milk chocolate was chosen because it is better tolerated compared to dark chocolate, has a more gentle profile of active ingredients (which can increase nausea and heartburn) and provides a source of available carbohydrates. The study will be conducted in accordance with the guidelines of the Ministry of Health's procedure for medical experiments on humans, and will be conducted after approval by the Institutional Helsinki Committee.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age ≥37 weeks
2. Single fetus in cephalic presentation
3. Spontaneous or induced labor in the active phase (dilation ≥ 5 cm).
4. Normal assessment of the mother and fetus upon admission to the delivery room (normal indices, normal monitoring and biophysical profile)
5. BMI 18-35 -

Exclusion Criteria:

1. Multiple pregnancies
2. Gestational age <37 weeks
3. Gestational or pre-gestational diabetes
4. Significant underlying diseases
5. Previous cesarean section/myomectomy
6. Known significant fetal malformation
7. Sensitivity to chocolate ingredients
8. Lack of documentation of necessary information -

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — It is limited due to the ability to give birth
Enrollment: 180 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Duration of second stage of labor | From full cervical dilation to delivery
  The duration of the second stage of labor, defined as the time in minutes from full cervical dulation (10cm) to delivery of the neonate.

SECONDARY OUTCOMES:
Mode of delivery | At delivery
  Mode of delivery categorized as spontanous vaginal delivery, operative vaginal delivery (vacuum), or cesarean delivery
Maternal nausea or vomiting during labor | From intervention administration untill discharge from labor room
  The occurrence of maternal nausea or vomiting during labor following the assigned intervention, as documented in the medical record
Neonatal Apgar score at 1 and 5 minutes | 1 and 5 minutes after delivery
  The Apgar score is assessed at 1 and 5 minutes after delivery. The total score ranges from 0 to 10, with higher scores indicating better neonatal condition.
Umbilical cord blood glucose level | at delivery
  Umbilical cord blood glucose concentration measured from umbelical blood collected immediately after delivery (when a cord blood sample is obtained per routine practice
Maternal heart rate | During the second stage of labor
  Maternal heart rate measured in beats per minute as recorded by continous intrapartum maternal monitorind
Umbelical cord blood PH | At delivery
  Umbelical cord blood PH measures immediatley after delivery

IPD SHARING:
Plan to Share IPD: No